CLINICAL TRIAL: NCT06378398
Title: An Early Phase 1 Trial of Omeprazole and Low Dose Aspirin to Identify Colorectal Biomarkers of Preventive Efficacy: The Omeprazole and Aspirin Polyp Prevention Study
Brief Title: A Trial of Omeprazole and Low Dose Aspirin to Identify Colorectal Biomarkers of Preventive Efficacy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UMCC 2023.037; HUM00247729 (Other: University of Michigan); UMI23-13-01 (Other: DCP Protocol Number); 1UG1CA242632-01A1 (NIH)
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasia
MeSH Terms: interventions — Omeprazole; Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention (Experimental): Two 20 mg/day omeprazole tablets and two 81 mg/day aspirin tablets taken before the first meal each day for 25-45 days.
  Interventions: Drug: Omeprazole; Drug: Aspirin

INTERVENTIONS:
Drug: Omeprazole — Two 20 mg/day omeprazole tablets taken before the first meal each day for 25-45 days.
  Other Names: Prilosec
Drug: Aspirin — Two 81 mg/day aspirin tablets taken before the first meal each day for 25-45 days.
  Other Names: Bayer Aspirin

SUMMARY:
This trial will obtain biomarker data on the possible preventive effects of omeprazole and low-dose aspirin in colorectal tissue. Persons who have had 5 or more adenomas, 5 or more serrated polyps, or an incompletely removed adenoma or serrated polyp in the colon or rectum are potentially eligible. Before participating in the study, study staff will explain the study and review the consent form. If you are interested and provide consent, study staff will then confirm your eligibility. Once enrolled, participants will take two 20 mg omeprazole tablets and two 81 mg aspirin tablets each day before the first meal each day for 25-45 days.

The study does involve biopsies of the colorectal tissue before and after taking the study medications. The biopsies are samples of tissue, about the size of a grain of rice, that will be taken from the colon or rectum before and after taking the study medications. This is done during a usual, clinical colonoscopy exam and during one more limited exam, called flexible sigmoidoscopy, that is done for the research study. The flexible sigmoidoscopy requires less preparation. Which procedure comes first depends on what fits best with each participant's clinical scenario. Biopsies of both normal mucosa and polyps (if possible) are collected.

DETAILED DESCRIPTION:
JAN2025 amendment added Adenomatous polyps meeting criteria for colon polyposis of unknown etiology (> 20 lifetime adenomas)

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Individuals who are due for a standard of care colonoscopy.
* Have a prior history of colorectal neoplasia including any ONE of the following:

  * Multiple (>=5) colorectal adenomas on most recent colonoscopy
  * Multiple (>=5) sessile serrated polyps on most recent colonoscopy
  * Adenomatous polyps meeting criteria for colon polyposis of unknown etiology (> 20 lifetime adenomas)
  * Serrated polyps meeting criteria for serrated polyposis syndrome
  * History of incompletely resected colorectal polyp(s) (adenoma or sessile serrated polyp) on most recent colonoscopy
* Willing to avoid taking non-steroidal anti-inflammatory drugs that are not provided by the study in the 30 days prior to Visit 1 and while on study.
* Willing to avoid taking proton pump inhibitors that are not provided by the study in the 30 days prior to Visit 1 and while on study.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation since endoscopy is not recommended during pregnancy.
* Demonstrate adequate organ and marrow function obtained within the last 60 days as defined below:

  * Absolute neutrophil count ≥1,000/microliter
  * Platelets ≥100,000/microliter
  * Total bilirubin ≤ 1.5 fold of the institutional upper limit of normal Note: Higher total bilirubin levels (≤ 3 mg/dL) can be allowed if due to known benign liver condition such as Gilbert's
  * AST (SGOT)/ALT (SGPT) ≤3.0 fold of the institutional upper limit of normal
  * Creatinine ≤1.5 fold of the institutional upper limit of normal
* Patients on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Age 76 or higher since there is an increased risk of GI bleeding and peptic ulcer disease in persons above 75 years of age.
* Pathogenic germline variants in adenomatous polyposis coli (APC) and DNA mismatch repair (MMR) genes associated with Lynch Syndrome, or biallelic pathogenic germline variants in the MutY homologue glycosylase (MUTYH) gene.
* Have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to proton pump inhibitors and/or aspirin.
* Participants may not be receiving any other investigational agents.
* Have a history of prior aspirin or NSAID gastritis with bleeding.
* Currently taking a proton pump inhibitor and unable/unwilling to discontinue use 30 days prior to Visit 1.
* Taking NSAIDs or aspirin >25% of the time (>8 days/month) and unable/unwilling to discontinue use 30 days prior to Visit 1 and until Visit 4.
* Currently taking medications associated with increased risk for bleeding (warfarin, Eliquis, Plavix, etc.).
* Currently taking medications that have interactions with omeprazole: atazanavir, erlotinib, levoketoconazole, nelfinavir, pazopanib, rilpivirine, sparsentan, certain azole antifungals (itraconazole, ketoconazole, and posaconazole).
* Have a history of hemophilia, Von Willebrand disease or any other known bleeding diathesis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Individuals who the site physician investigator assesses as at high risk for bleeding due to heavy alcohol use or comorbid conditions.
* Pregnant women are excluded since endoscopy is not recommended while pregnant.
* Have invasive cancer or being treated for invasive cancer at the current time or within the past 36 months, with the exception of cancers curatively removed by surgery, other than melanoma, and stage I and II cervical squamous cell cancers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Identification of biomarkers for omeprazole/aspirin combination treatment in the human colorectum | up to 45 days from intervention initiation
  The ratio of Ki67 proliferation marker to cleaved caspase 3 apoptosis marker, and changes in gene expression by high throughput RNA sequencing (RNA-Seq).

SECONDARY OUTCOMES:
Evaluation of gene expression changes | up to 45 days from intervention initiation
  To compare gene expression changes by RNA-Seq observed in the clinical trial with that observed in a well-characterized rodent colon cancer prevention model to evaluate potential for preventive efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Zora Djuric, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - The University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared